CLINICAL TRIAL: NCT07070713
Title: Assess and Compare the Efficacy and Safety of FOLFOX Combined With Cetuximab Versus FOLFOXIRI Combined With Bevacizumab When Both Used in Combination With QL1706 for First-line Treatment of Metastatic Colorectal Cancer With Left-sided Primary Tumors.
Brief Title: Efficacy and Safety of FOLFOX+Cetuximab vs. FOLFOXIRI+Bevacizumab Both With QL1706 in First-Line Treatment of Left-Sided mCRC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYLT-031
Record Dates: First submitted 2025-07-09; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Colorectal Cancer With Left-sided Primary Tumor; Immunotherapy
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group：FOLFOXIRI + QL1706 + Bevacizumab (Experimental): FOLFOXIRI (irinotecan 165 mg/m², iv, d1; oxaliplatin 85 mg/m², iv, d1; (levo)leucovorin 400 mg/m², iv, d1; 5-FU total dose 2400 mg/m², iv infusion (continuous for 48 hours), d1) +QL1706 (5mg/kg, i.v, Q3W) + bevacizumab (5 mg/kg, i.v., every 2 weeks).
  Interventions: Drug: FOLFOXIRI + QL1706 + Bevacizumab
- B group：FOLFOX + QL1706 + Cetuximab (Active Comparator): FOLFOX (oxaliplatin 85 mg/m², intravenous infusion (2 hours), day 1; (levo)leucovorin (200) 400 mg/m², intravenous infusion (2 hours), day 1; 5-FU 400 mg/m², intravenous injection, followed by 2400 mg/m², intravenous infusion (continuous for 46-48 hours), day 1) +QL1706 (5mg/kg, i.v, Q3W) + cetuximab (500 mg/m², intravenous infusion, every 2 weeks).
  Interventions: Drug: FOLFOX+QL1706+Cetuximab

INTERVENTIONS:
Drug: FOLFOXIRI + QL1706 + Bevacizumab — FOLFOXIRI(Irinotecan 165mg/m², iv, d1; Oxaliplatin 85mg/m², iv, d1; (Levo) Folinic Acid (200) 400mg/m², iv, d1; total 5-FU 2400mg/m², iv gtt (continuous for 48h), d1) + QL1706 (5mg/kg, i.v., Q3W) + Bevacizumab (5mg/kg, i.v., Q2W)
  Arms: A group：FOLFOXIRI + QL1706 + Bevacizumab
Drug: FOLFOX+QL1706+Cetuximab — FOLFOX (Oxaliplatin 85mg/m², iv gtt (for 2h), d1; (Levo) Folinic Acid (200) 400mg/m², iv gtt (for 2h), d1; 5-FU 400mg/m², iv, followed by 2400mg/m², iv gtt (continuous for 46-48h), d1) + QL1706 (5mg/kg, i.v., Q3W) + Cetuximab (500mg/m², i.v., Q2W).
  Arms: B group：FOLFOX + QL1706 + Cetuximab

SUMMARY:
This is a two-arm, randomized phase II clinical study. It is planned to enroll 44 patients with primary left-sided, RAS and BRAF wild-type metastatic colorectal cancer. After signing the informed consent, eligible subjects will be screened to enter the clinical study and assigned to two treatment groups using simple randomization and allocation concealment methods.

The treatment plans for the two groups are as follows:

Group A: FOLFOXIRI (Irinotecan 165mg/m², iv, d1; Oxaliplatin 85mg/m², iv, d1; (Levo) Folinic Acid (200) 400mg/m², iv, d1; total 5-FU 2400mg/m², iv gtt (continuous for 48h), d1) + Bevacizumab (5mg/kg, i.v, Q2W) Group B: FOLFOX (Oxaliplatin 85mg/m², iv gtt (for 2h), d1; (Levo) Folinic Acid (200) 400mg/m², iv gtt (for 2h), d1; 5-FU 400mg/m², iv, followed by 2400mg/m², iv gtt (continuous for 46-48h), d1) + Cetuximab (500mg/m², i.v, Q2W) Both groups A and B will repeat the treatment every 2 weeks, for a maximum of 9 cycles. Then, the attending physician will decide whether to conduct maintenance treatment (Capecitabine or 5FU/LV with or without Bevacizumab is recommended).

Both groups A and B will be combined with QL1706 (5mg/kg, i.v, Q3W) for a maximum of 52 weeks.

Medication will continue until the researcher judges that there is no longer clinical benefit (the researcher makes a comprehensive judgment based on RECIST v1.1 imaging evaluation and clinical status, etc.), intolerable toxicity occurs, the subject withdraws informed consent, or other criteria for terminating treatment in the protocol are met, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old.
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
3. Histologically or cytologically confirmed metastatic colorectal adenocarcinoma with the primary tumor located in the left-sided colon (from the splenic flexure to the rectum), including cecal adenocarcinoma.
4. Presence of at least one evaluable lesion according to RECIST v1.1 criteria.
5. The subject has provided sufficient tumor tissue samples through colonoscopy biopsy for MSI, TMB, and other tests.
6. Tumors confirmed by tissue testing to be wild-type for KRAS, NRAS, and BRAF.
7. Within 7 days prior to the first dose of study drug, laboratory tests meet the following criteria (no blood products, hematopoietic growth factors, albumin, or other corrective treatments within 14 days prior to testing): (1) Biochemistry: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal (ULN), or ≤ 5 times ULN in the presence of liver metastases; total bilirubin (TBIL) ≤ 1.5 times ULN, or ≤ 2 times ULN in the presence of liver metastases; serum creatinine ≤ 1.5 times ULN, or creatinine clearance > 50 mL/min (calculated by the Cockcroft-Gault formula). (2) Hematology: Hemoglobin (Hb) ≥ 9.0 g/dL. No red blood cell transfusions within 1 week prior to the baseline Hb test; absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; platelet count ≥ 100 × 10⁹/L. No platelet transfusions within 1 week prior to the baseline platelet test. (3) Coagulation function: International normalized ratio (INR) ≤ 1.5 × ULN (for subjects receiving prophylactic anticoagulation therapy without active bleeding [i.e., no bleeding within the past 14 days], the investigator should determine that the INR is within a safe and effective therapeutic range). (4) Urinalysis: Urine protein ≤ 30 mg/dL (1+) by dipstick or routine urinalysis (if ≥ 2+, then a 24-hour urine protein quantification must be < 1 g/24h).
8. Estimated survival of at least 3 months.
9. No contraindications to chemotherapy or immunotherapy.
10. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment and agree to use a reliable and effective method of contraception during the study and for 5 months after the last dose of study drug. Men whose partners are women of childbearing potential must agree to use a reliable and effective method of contraception during the study and for 5 months after the last dose of study drug. Lactating women are not eligible.
11. The subject must provide informed consent for the study prior to enrollment, voluntarily sign a written informed consent form, and be willing and able to comply with the study visit schedule, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Confirmed by histopathological or cytological examination as other pathological types, such as squamous cell carcinoma, undifferentiated carcinoma, neuroendocrine carcinoma, etc. For mixed pathological types, the determination will be made based on the predominant component; adenocarcinoma component > 70% confirmed by pathologist is eligible for enrollment. Primary appendiceal tumors are exclusion criteria.
2. Presence of other active malignancies within the past 3 years, except for early malignancies that have been cured (carcinoma in situ or stage I tumors), such as adequately treated cervical carcinoma in situ, thyroid cancer, basal cell or squamous cell carcinoma of the skin, etc.
3. Previous systemic therapy for unresectable/metastatic colorectal cancer.
4. Active autoimmune disease within the past 2 years requiring systemic treatment (i.e., immunomodulatory drugs, corticosteroids, or immunosuppressive agents); however, replacement therapy (e.g., thyroid hormone, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) will not be considered systemic treatment and is permitted.
5. Presence of immunodeficiency or receipt of long-term systemic corticosteroid therapy (daily dose > 10 mg prednisone or equivalent corticosteroid) within 7 days prior to enrollment, or other immunosuppressive therapy.
6. Uncontrolled diabetes mellitus; peripheral neuropathy ≥ Grade 2.
7. Active tuberculosis, or receipt of anti-tuberculosis treatment within 1 year prior to enrollment.
8. If hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) are positive, the patient's HBV-DNA must be less than 500 IU/mL. For patients with active hepatitis B, the patient must have received antiviral therapy for at least 14 days prior to enrollment (according to local standard treatment, such as entecavir or tenofovir) and agree to continue effective antiviral therapy during the study.
9. If HCV antibody is positive, HCV-RNA testing will be performed; if HCV-RNA > 1,000 copies/mL, the patient will be excluded.
10. Receipt of any live vaccine within 28 days prior to enrollment (e.g., vaccines for infectious diseases, such as influenza vaccine, varicella vaccine, etc.).
11. Previous allogeneic bone marrow transplant or solid organ transplant.
12. Major surgery within 4 weeks prior to the first dose, or significant trauma, or presence of a wound that has not healed or healed poorly or complications in wound management.
13. Known allergy to any component of the study drug; known multiple allergies or history of severe allergic diseases.
14. Systemic anti-infective therapy within 2 weeks prior to the first dose.
15. Receipt of nonsteroidal anti-inflammatory drugs, antiplatelet agents, or anticoagulants within 7 days prior to the first dose or ongoing.
16. Active infectious diseases, such as HIV/AIDS or active syphilis.
17. Use of any other investigational drug within 28 days prior to randomization or participation in another investigational drug trial.
18. Clinically significant underlying medical conditions that may affect the administration of the study drug or compliance with the protocol, as judged by the investigator.
19. Known history of psychiatric illness, drug abuse, alcoholism, or drug addiction.
20. Pregnant or breastfeeding women.
21. Other individuals deemed inappropriate for enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 18 weeks
  The percentage of participants in the analysis dataset who achieve a best overall response of Complete Response (CR) or Partial Response (PR) from the start of treatment until disease progression or withdrawal from the study.

SECONDARY OUTCOMES:
Duration of Response | 52 weeks
  The time from the first assessment of Complete Response (CR) or Partial Response (PR) until the first assessment of Progressive Disease (PD) or death from any cause.
Disease Control Rate | 18 weeks
  The proportion of patients whose tumors have shrunk or remained stable for a certain period of time, including cases of Complete Response (CR), Partial Response (PR), and Stable Disease (SD).
Progression Free Survival | 52 weeks
  The time from the day of enrollment until the first occurrence of disease progression (PD) or death due to any cause.
Overall Survival | 52 weeks
  It refers to the time from the date of enrollment to the date of death due to any cause.
Incidence of Adverse Events | 30 days after the end of study
  fatigue, nausea/vomiting, abdominal pain and diarrhea, stomatitis, hepatic dysfunction, myelosuppression, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No